CLINICAL TRIAL: NCT06255756
Title: Effect of Acupuncture Therapy on Dysphagic Parkinson's Patients: A Randomized Controlled Study
Brief Title: Effect of Acupuncture Therapy on Dysphagic Parkinson's Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: ethical issues
Sponsor: Zeng Changhao (Other)
Responsible Party: Sponsor-Investigator, Zeng Changhao, Research Director, People's Hospital of Zhengzhou University
Organization: People's Hospital of Zhengzhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Zhenjiu-Parkinson
Record Dates: First submitted 2024-02-04; First posted 2024-02-13 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Dysphagia
MeSH Terms: conditions — Deglutition Disorders | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- routine treatment+swallowing rehabilitation training+acupuncture therapy (Experimental): The experimental group was given routine treatment and swallowing rehabilitation training. Moreover, the experimental group was given acupuncture therapy.
  Interventions: Behavioral: Routine rehabilitation training; Behavioral: Swallowing rehabilitation training; Procedure: Acupuncture therapy
- routine treatment+swallowing rehabilitation training (Active Comparator): The control group was given routine treatment and swallowing rehabilitation training.
  Interventions: Behavioral: Routine rehabilitation training; Behavioral: Swallowing rehabilitation training

INTERVENTIONS:
Behavioral: Routine rehabilitation training — Balance function training: Patients were instructed to achieve weight shift between the left and right sides of the balance bar in a standing position.
  Walking function training: based on hip, knee, and ankle control training, patients were instructed to take steps training.
  Core muscle strength training: Patients were instructed to maintain 3 minutes of training in Bridge-style movement.
  Functional training of daily living: including training on dressing and undressing, independent eating, painting, and writing.
  Routine rehabilitation training was performed 30-45 minutes/time, 1-2 times/day, 5-7 days/week.
Behavioral: Swallowing rehabilitation training — Swallowing-related organ training involves various exercises targeting the lip, mandibular muscle, cheek, tongue muscle, soft palate, as well as exercises for vocal cord closure, laryngeal lifting, and pharyngeal muscle training. These exercises are performed for 5-15 minutes each session, 1-2 times per day, and 5-7 days per week.
  Sensory stimulation training is conducted using a self-made popsicle, where medical staff gently stimulate the patient's cheek, palatoquadrate, soft palate, posterior pharyngeal wall, tongue surface, and sublingual area repeatedly. Each session lasts 5-25 minutes, performed 1-3 times per day, and 3-7 days per week.
  Once the patient's swallowing function improves to a certain extent, allowing for safe oral intake, direct training or oral feeding training can be gradually introduced.
Procedure: Acupuncture therapy — The whole acupuncture therapy was performed once daily for 5 days per week, including acupuncture needle and tongue needle.
  Acupuncture needle:
  Main acupoints: Lianquan, Shanglianquan (depression between the hyoid bone and the lower border of the mandible), Yifeng; Auxiliary acupoints: Fengchi, Wangu, Fengfu, Yamen, Neidaying (depression of 1 inch below the anterior margin of the mandible).
  Tongue needle (pricking):
  Acupoints: Jinjin, Yuye, posterior pharyngeal wall (both sides of the uvula).
  Arms: routine treatment+swallowing rehabilitation training+acupuncture therapy

SUMMARY:
We are currently conducting a randomized controlled study in China, specifically in three hospitals' rehabilitation medicine departments, focusing on dysphagic participants with Parkinson's disease. The aim of our study is to evaluate the effectiveness of acupuncture therapy as an additional intervention for these participants. Participants were randomly assigned to either the experimental group or the control group, with 56 individuals in each group. Both groups are receiving standard treatment and swallowing rehabilitation training, while the experimental group is also receiving acupuncture therapy. Our study aims to provide valuable insights into the potential benefits of acupuncture in improving swallowing difficulties in Parkinson's disease participants.

DETAILED DESCRIPTION:
We are currently conducting a randomized controlled study in China, specifically in three hospitals' rehabilitation medicine departments, focusing on dysphagic participants with Parkinson's disease. The aim of our study is to evaluate the effectiveness of acupuncture therapy as an additional intervention for these participants. Participants were randomly assigned to either the experimental group or the control group, with 56 individuals in each group. Both groups are receiving standard treatment and swallowing rehabilitation training, while the experimental group is also receiving acupuncture therapy. Our study aims to provide valuable insights into the potential benefits of acupuncture in improving swallowing difficulties in Parkinson's disease participants.

The study lasted 42 days (6 weeks) for each participant. Specifically, our main focus is on the study of Lianquan, Shanglianquan (depression between the hyoid bone and the lower border of the mandible), Yifeng, Fengchi, Wangu, Fengfu, Yamen, Neidaying (depression of 1 inch below the anterior margin of the mandible), Jinjin, Yuye, posterior pharyngeal wall (both sides of the uvula).

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years.
* Meeting the diagnostic criteria for Parkinson's disease.
* Diagnosed with dysphagia confirmed by the video fluoroscopic swallowing study.
* Water swallow test> Level 3.
* Stable vital signs, conscious, able to cooperate with assessment and treatment.

Exclusion Criteria:

* Dysphagia possibly caused by other reasons, such as cerebrovascular disease, trauma, neuromuscular diseases, malignant diseases of the pharynx and larynx, and digestive tract diseases.
* History of mental diseases or use of antipsychotics.
* Complicated with cognitive impairment or consciousness dysfunction.
* Simultaneously suffering from severe liver, kidney failure, tumors, or hematological diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Penetration-Aspiration Scale-liquid | Day 1 and Day 42
  The Penetration-Aspiration Scale (PAS) was conducted under video fluoroscopic swallowing study. PAS is a standardized tool used to assess the safety of swallowing. The scale was developed to evaluate the entry of material into the airway (penetration) and the subsequent passage of material below the vocal folds (aspiration) during swallowing. The PAS scale ranges from 1 to 8, with each level representing different degrees of penetration or aspiration.
  In this assessment, we used 60% barium sulfate suspension A higher level of PAS indicated a severer dysphagia.
Penetration-Aspiration Scale-paste | Day 1 and Day 42
  The Penetration-Aspiration Scale (PAS) was conducted under video fluoroscopic swallowing study. PAS is a standardized tool used to assess the safety of swallowing. The scale was developed to evaluate the entry of material into the airway (penetration) and the subsequent passage of material below the vocal folds (aspiration) during swallowing. The PAS scale ranges from 1 to 8, with each level representing different degrees of penetration or aspiration.
  In this assessment, we used 180% barium sulfate suspension A higher level of PAS indicated a severer dysphagia.

SECONDARY OUTCOMES:
Swallowing time | Day 1 and Day 42
  The assessment was conducted under video fluoroscopic swallowing study. A 60% barium sulfate suspension was mixed with different doses of thickening agents. The liquid (60% barium sulfate suspension) was used. A shorter time indicated better swallowing function.
body mass index | Day 1 and Day 42
  Patients' body mass index was assessed with the physical check, with the combination of height and body weight. as kg/m^2, reference range: 18.5 kg/m2≤BMI<24 kg/m2.
Serum Albumin | Day 1 and Day 42
  Patients' Serum Albumin was assessed from the routine blood test, reference range: 35~50 g/L.Values below the reference range for these indicators indicated an unsatisfying nutritional status (risk of malnutrition).
Prealbumin | Day 1 and Day 42
  Patients' Prealbumin was assessed from the routine blood test, reference range: 200~400 mg/L.Values below the reference range for these indicators indicated an unsatisfying nutritional status (risk of malnutrition).
Hemoglobin | Day 1 and Day 42
  Patients' Hemoglobin was assessed from the routine blood test, reference range: males: 120~160 g/L, females: 110~150 g/L. Values below the reference range for these indicators indicated an unsatisfying nutritional status (risk of malnutrition).
Swallowing Quality of Life | Day 1 and Day 42
  Swallowing Quality of Life (SWAL-QOL) is a questionnaire designed to evaluate the impact of swallowing problems on a patient's quality of life. It includes 44 items covering various aspects such as eating desire, food selection, communication, and mental health.
  The SWAL-QOL total score ranges from 0 to 100, with higher scores indicating better quality of life. Therefore, in this case, the higher the score, the better the individual's quality of life related to their swallowing function.

CONTACTS AND LOCATIONS:
Overall Officials: Nieto Luis, Master, Study Director — Site Coordinator of United Medical Group
Locations (1):
- Zheng Da yi Yuan Hospital, Zhenzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No